CLINICAL TRIAL: NCT04748679
Title: Cognitive Behavioral Therapy (CBT) Study Evaluating the Updating of Persecutory Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Julia Sheffield, Assistant Professor of Psychiatry & Behavioral Sciences, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201882
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Psychosis; Persecutory Delusion
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Worry Intervention (Experimental): The Worry Intervention uses cognitive-behavioral therapy (CBT) techniques to support the patient in reducing the amount of time they worry throughout the week. It is an 8-week manualized treatment with 5 modules. Each session is 45-60 minutes.
  Interventions: Behavioral: Worry Intervention
- Befriending (Active Comparator): Befriending therapy controls for the general factors of therapy (warmth, engagement) without any 'active' interventions. Individuals in the befriending arm will spend sessions talking with the therapist about things that interest them. It will also be conducted over 8-weeks with 45-60 minute sessions.
  Interventions: Behavioral: Befriending

INTERVENTIONS:
Behavioral: Worry Intervention — The worry intervention is weekly individual therapy with a trained therapist
  Arms: Worry Intervention
Behavioral: Befriending — The worry intervention is weekly individual therapy with a trained therapist
  Arms: Befriending

SUMMARY:
The purpose of this study is to examine how Bayesian belief updating changes throughout psychotherapeutic treatment for persecutory delusions. Specifically, individuals with a psychotic disorder diagnosis who endorse both a current persecutory delusion with strong conviction and significant worry will be recruited and randomized to receive either a CBT-based worry intervention for persecutory delusions or an active control condition (befriending therapy). The investigators will examine: 1) whether belief updating parameters change as delusion severity changes, 2) whether CBT contributes to greater change in belief updating parameters than befriending therapy, and 3) whether neural correlates of belief updating parameters, as measured using functional magnetic resonance imaging (fMRI), predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 - 65.
2. Communicative in English.
3. Premorbid Intelligence >79 (WTAR)
4. Provide voluntary, written informed consent.
5. Physically healthy by medical history.
6. Weight <300 lbs
7. Stable medication regimen over at least the past two weeks, including the use of either an oral or intramuscular administration of an antipsychotic medication.
8. Diagnosis of a non-affective psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, brief psychotic disorder, psychosis NOS) confirmed by Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-5 (SCID) or diagnostic interview with a trained clinician.
9. A persecutory delusion scoring at least a 3 on the conviction scale of the Psychotic Symptoms Rating Scale (PSYRATS) that had persisted for at least two weeks and that was not considered the direct result of substance use
10. A clinically significant level of worry, as shown by a score of at least 44 on the Penn State Worry Questionnaire (PSWQ).

Exclusion Criteria:

1. Age less than 18 or greater than 65.
2. Not communicative in English.
3. Premorbid IQ < 79 (WTAR)
4. Unable to provide written informed consent.
5. Current medical or neurological illness.
6. History of severe head trauma.
7. Weight >300 lbs
8. Primary diagnosis of alcohol or substance use disorder or personality disorder
9. Conditions that preclude fMRI scanning (as defined in the fMRI Screening Form)
10. Subjects who are actively involved with individual cognitive therapy (Past experience with individual therapy is not an exclusion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Computational Parameters of Belief Updating as Measured During a Probabilistic Reversal Learning Task | Baseline, 4 weeks, 8 weeks, 24 weeks
  change in computational parameters after intervention
Change in Delusion Severity Utilizing the Change in Psychotic Symptoms Rating Scale (PSYRATS) | Baseline, 4 weeks, 8 weeks, 24 weeks
  The change in the Delusions subscale total of the Psychotic Symptoms Rating Scale (PSYRATS) from Baseline to Week 24. The Delusions subscale is a composite score of 6 items each rated from 0-4 with 4 indicating more severe symptomology. The Delusions subscale has a possible range of 0-24.
Change in Neural Correlates of Belief Updating Parameters | Baseline, 8 weeks
  Change in blood oxygen dependent level (BOLD) signal after intervention

SECONDARY OUTCOMES:
Baseline Neural Predictors of Treatment Response | Baseline
  BOLD signal during belief updating task at baseline predicting treatment response
Resting-State Predictors of Treatment Response | Baseline
  resting-state connectivity of functional networks predicting treatment response

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheffield JM, Sloan AF, Corlett PR, Rogers BP, Vandekar S, Liu J, Beals KM, Hall LM, Gautier T, Moussa-Tooks AB, Torregrossa LJ, Achee M, Armstrong K, Woodward ND, Belt K, Freeman D, Isham L, Diamond R, Brinen AP, Heckers S. Prior Expectations of Volatility Following Psychotherapy for Delusions: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2517132. doi: 10.1001/jamanetworkopen.2025.17132. PMID 40553472